CLINICAL TRIAL: NCT03669783
Title: Randomized Open-label Non-inferiority Phase 3 Clinical Trial for Patients With a Stage IV Childhood Renal Tumor, Comparing Upfront Vincristine, Actinomycin-D and Doxorubicin (Standard Arm) With Upfront Vincristine, Carboplatin and Etoposide (Experimental Arm)
Brief Title: Clinical Trial for Patients With a Stage IV Childhood Renal Tumor, Comparing Upfront Vincristine, Actinomycin-D and Doxorubicin (Standard Arm) With Upfront Vincristine, Carboplatin and Etoposide (Experimental Arm)
Acronym: RANDOMET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-07
Record Dates: First submitted 2018-08-27; First posted 2018-09-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Childhood Renal Tumor
MeSH Terms: interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment VAD (Active Comparator): Vincristin, Actinomycin-D and Doxorubicin
  Interventions: Drug: treatment Vincristin; Drug: treatment Actinomycin-D; Drug: treatment Doxorubicin
- treatment VCE (Experimental): Vincristin, Carboplatin and Etoposide
  Interventions: Drug: treatment Vincristin; Drug: treatment Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: treatment Vincristin — 1 x Vincristin 1,5mg/m² iv bolus day 1 in week 1,2,3,4,5,6
Drug: treatment Actinomycin-D — 1 x Actinomycin D 45µg/kg iv bolus day 1 in week 1, 3, 5
  Arms: treatment VAD
Drug: treatment Doxorubicin — 1 x Doxorubicin 50mg/m² 6h Infusion day 1 in week 1,5
  Arms: treatment VAD
Drug: treatment Carboplatin — 1 x Carboplatin 200 mg/m² 1h infusion day 1,2,3 in week 1,4
  Arms: treatment VCE
Drug: Etoposide — 1 x Etoposide 100mg/m² 1h infusion day 1,2,3 in week 1,4
  Arms: treatment VCE

SUMMARY:
Nephroblastoma (Wilms tumor, WT) is the most common renal tumor of childhood representing ± 6% of all childhood malignancies. The diagnosis is established on clinical and radiological grounds. Metastases are visible on conventional imaging in at least 12% of nephroblastoma patients; however, an additional ~15% of patients have nodules on CT-scan only. The treatment consists of neoadjuvant (preoperative) chemotherapy, nephrectomy and risk-based adjuvant chemotherapy ± radiation therapy (RT) to the flank and/or metastases. For truly localized tumors, overall survival is > 85% (high risk histology excluded). Several high risk biological characteristics have been identified: diffuse anaplasia, gain of 1q chromosome, loss of heterozygosity 1p + 16q, blastemal residual volume.

For metastatic nephroblastoma, the standard neo-adjuvant chemotherapy includes 3 drugs: vincristine, actinomycin-D and doxorubicin (VAD). Long-term survival is 82% (1). However, two issues arise. First, the use of doxorubicin ± concomitant RT might be associated with cardiac and pulmonary sequelae (4-17% of congestive heart failure) (2), and actinomycin-D is associated with hepatic toxicity (3). Second, patients with "CT-only" nodules are treated according to "localized disease". However, their outcome is poorer than that of truly "localized disease" (4-6).

The efficacy of carboplatin and etoposide is known for a long time; these drugs are used as second line treatment or for high-risk histology nephroblastoma. Therefore, an alternate chemotherapy has been designed that combines drugs shown as highly efficacious in nephroblastoma, i.e., Vincristine, Carboplatin and Etoposide (VCE). VCE has been used for the treatment of other pediatric malignancies. For metastatic nephroblastoma, the switch from VAD to VCE and the associated reduction of actinomycin-D and doxorubicin is expected to reduce the chemotherapy-related long-term toxicity. In addition, VCE could potentially decrease the rate of patients requiring pulmonary RT. Finally VCE may have a beneficial effect on tumor high risk biological characteristics.

French patients with nephroblastoma have been treated for > 40 years according to SIOP protocols collaborating in the SIOP Renal Tumour Study Group (SIOP-RTSG). This group has designed an international randomized phase III clinical trial for the evaluation of VCE versus VAD in patients with metastatic renal tumors (>>90% having nephroblastoma), in order to decrease the long-term toxicity while at least preserving, if not improving, the treatment efficacy. In addition, the issue of "CT-only" nodules and their adequate treatment needs to be solved. In previous protocols, the treatment strategy was based on the diagnosis of pulmonary metastases (~90% of all metastases) by conventional pulmonary X-ray. Central Radiological Review (CRR) is planned for the initial staging using CT ± MRI, as it is expected to more accurately detect patients with metastatic disease, including patients with "CT-only" nodules. In addition, CRR will be set up for real-time response assessment during treatment, in order to reliably determine who require pulmonary RT and which postoperative chemotherapy.

Therefore, the main trial objectives are:

* Explore the non-inferiority (efficacy) of neoadjuvant VCE chemotherapy (experimental arm) as compared to the standard arm with VAD.
* Provide central radiological review (CRR) at diagnosis and after neoadjuvant chemotherapy in order to determine more precisely the appropriate treatment for each patient.

The primary objective of the RCT is to investigate the metastatic complete response rate (MetCR, including very good partial response (VGPR)) of neoadjuvant 6 weeks of VAD as compared to neoadjuvant VCE in stage IV renal tumours using CRR. Several international studies have shown that MetCR is a good surrogate endpoint for survival.

The postoperative treatment, secondary objectives as well as the intended methodology are detailed in the research project.

The total number of patients is 406 patients for the entire phase III trial running in the 12 major SIOP countries (max 110 patients in France).

The expected trial duration is 5 years for accrual + 2 years follow-up (the overall 10-year follow-up for long-term toxicity will be an independently funded ancillary study. This duration is required for a reliable evaluation of the cardiac toxicity).

The results of the current trial should be useful for the future protocols for the treatment of all patients with nephroblastoma (metastatic but also localized and bilateral).

The results of this RCT will be worthy for the entire international pediatric oncology community and future patients throughout the world and will be communicated in scientific congresses and high-level peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* suffering from metastatic renal tumour at initial diagnosis
* having at least one circumscript, non-calcified (pulmonary) nodule (or other lesion highly suspicious of metastasis according to criteria for metastatic disease) ≥ 3 mm as determined by chest CT-scan and abdominal CT-scan/MRI.
* Metastatic disease must be confirmed by central review.

Exclusion Criteria:

-

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2028-10-03 (Estimated); Study Completion 2033-10-03 (Estimated)

PRIMARY OUTCOMES:
Metastatic response assessment by neoadjuvant chemotherapy only | 6 weeks
  percentage of patients with complete response (CR) or Very Good Partial Response (VGPR) of metastasis of nephroblastoma after 6 weeks of preoperative chemotherapy

SECONDARY OUTCOMES:
Secondary metastatic response assessment | 6 weeks
  percentage of patients after 6 weeks of preoperative chemotherapy achieving a CR after surgery of metastasis at time of nephrectomy
Clinical outcome after treatment | 2 and 5 years
  stage of local tumor (for each arm)
Histological response to preoperative treatment | 6 weeks
  stage distribution of local tumor histological subtype distribution of local tumor (low, intermediate or high risk (LR, IR, HR))

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO-PRADALIE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No